CLINICAL TRIAL: NCT04550884
Title: Neuropathic Foot and Ankle in Rheumatoid Arthritis : Ultrasound and Nerve Conduction Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Taher Mohamed Amin, principal investigator, Assiut University
Other Study IDs: neuropathic foot and ankle
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: neuromascular ultrasound — neuromascular ultrasound of foot and ankle
  Other Names: nerve conduction study

SUMMARY:
1. To measure the prevalence of Neuropathic pain in Rheumatoid arthritis patients with ankle and foot pain
2. To evaluate the role of Neuromuscular Ultra sound (NMUS) and nerve conduction study (NCS) in assessment of Neuropathic foot and ankle in Rheumatoid arthritis patients

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common chronic systemic autoimmune disease that primarily affects the lining of the synovial joints which symmetrically involves the small joints, can cause cartilage and bone damage and associated with progressive disability, premature deaths, and socioeconomic burdens .

In RA, neuropathic pain "which is defined as pain caused by a lesion or a disease of the somatosensory system" , could be suggested by :nerve compression, associated comorbidities and vascuilitis .

Despite the recent advancement in RA treatment, neuropathic pain remains a cause of persistent pain even in controlled disease activity.

The prevalence of clinical neuropathy varies from 0.5% to 85% in patients with RA, which can cause functional disability . Foot and ankle pain is highly prevalent in RA with peripheral neuropathy is a common contributor to it . In previous studies , it was found that the most foot neuropathies are of tarsal tunnel syndrome, peroneal nerve entrapment and pure sensory axonal neuropathy.

For evaluation of neuropathic foot and ankle in RA , electrophysiological and imaging techniques can be very useful.

Nerve conduction study (NCS) is the electrodiagnostic evaluation of the function of peripheral nerves ,it can provide information regarding the presence, severity and location of a lesion, symmetricity of neuropathy, mononeuropathy or disorders affecting the neuromuscular junctions. Also, the functional modality most involved (sensory or motor) and the predominant pattern of pathology (e.g., axonal, demyelinating, or both.

Neuromascular ultrasond(NMUS) is a new modality of diagnosis developed in the past 20 years , and it can assess anatomical abnormalities that can't be evaluated by NCS NMUS being noninvasive and inexpensive diagnostic modality , it has been introduced as a complement to NCS for diagnosis of nerve conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years.
2. RA patients who fulfilled the 2010 ACR/European league against Rheumatism(EULAR) criteria for the classification of RA
3. RA patients complaining of foot and ankle pain

Exclusion Criteria:

1. Presence of other autoimmune disorders
2. Presence of any comorbidities causing neuropathy as Diabetes Mellitus, disc prolapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients with foot and ankle pain attending at both inpatient department and outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
ultrasound parameters | 3 years
  nerve cross-section

SECONDARY OUTCOMES:
nerve conduction parameters | 3 years
  nerve distal latency
painDETECT questionnaire | 1 year
  screening for neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: EMAN A AL Kady, professor, Study Director — Assiut University

REFERENCES:
- [Background] Abu-Shaheen A, Yousef S, Riaz M, Nofal A, AlFayyad I, Khan S, Heena H. Testing the validity and reliability of the Arabic version of the painDETECT questionnaire in the assessment of neuropathic pain. PLoS One. 2018 Apr 23;13(4):e0194358. doi: 10.1371/journal.pone.0194358. eCollection 2018. PMID 29684014
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Aseem F, Williams JW, Walker FO, Cartwright MS. Neuromuscular ultrasound in patients with carpal tunnel syndrome and normal nerve conduction studies. Muscle Nerve. 2017 Jun;55(6):913-915. doi: 10.1002/mus.25462. Epub 2016 Nov 18. PMID 27859374
- [Background] Colloca L, Ludman T, Bouhassira D, Baron R, Dickenson AH, Yarnitsky D, Freeman R, Truini A, Attal N, Finnerup NB, Eccleston C, Kalso E, Bennett DL, Dworkin RH, Raja SN. Neuropathic pain. Nat Rev Dis Primers. 2017 Feb 16;3:17002. doi: 10.1038/nrdp.2017.2. PMID 28205574
- [Background] El-Hewala, A. E.-S., Soliman, S., Labeeb, A., Zytoon, A. and El-Shanawany, A. (2016) 'Foot neuropathy in rheumatoid arthritis patients: clinical, electrophysiological, and ultrasound studies', Egyptian Rheumatology and Rehabilitation. Springer Science and Business Media LLC, 43(3), p. 85. doi: 10.4103/1110-161x.189640.
- [Background] Fransen J, van Riel PL. The Disease Activity Score and the EULAR response criteria. Rheum Dis Clin North Am. 2009 Nov;35(4):745-57, vii-viii. doi: 10.1016/j.rdc.2009.10.001. PMID 19962619
- [Background] Kaeley N, Ahmad S, Pathania M, Kakkar R. Prevalence and patterns of peripheral neuropathy in patients of rheumatoid arthritis. J Family Med Prim Care. 2019 Jan;8(1):22-26. doi: 10.4103/jfmpc.jfmpc_260_18. PMID 30911476
- [Background] Ten Klooster PM, de Graaf N, Vonkeman HE. Association between pain phenotype and disease activity in rheumatoid arthritis patients: a non-interventional, longitudinal cohort study. Arthritis Res Ther. 2019 Nov 29;21(1):257. doi: 10.1186/s13075-019-2042-4. PMID 31783899
- [Background] Koop SM, ten Klooster PM, Vonkeman HE, Steunebrink LM, van de Laar MA. Neuropathic-like pain features and cross-sectional associations in rheumatoid arthritis. Arthritis Res Ther. 2015 Sep 3;17(1):237. doi: 10.1186/s13075-015-0761-8. PMID 26335941
- [Background] McWilliams DF, Walsh DA. Pain mechanisms in rheumatoid arthritis. Clin Exp Rheumatol. 2017 Sep-Oct;35 Suppl 107(5):94-101. Epub 2017 Sep 29. PMID 28967354